CLINICAL TRIAL: NCT04415788
Title: Novel Versus Traditional Inspiratory Muscle Training Regimens as Home-based, Stand-alone Therapies in COPD
Brief Title: Inspiratory Muscle Training and COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ladislav Batalik, Principal investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BrnoUH RHO AZVj 2021
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Pulmonary rehabilitation; Telemedicine; Quality of life; Inspiratory muscle training; Test of incremental respiratory endurance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test of Incremental Respiratory Endurance - IMT (Experimental): Training will consist of six levels (A-F) with six inspirations at each level for up to 36 breaths per session. TIRE data will be stored in the tablet and automatically synced to account on cloud-based online platform for subsequent interrogation and data retrieval. Before every training session, subjects will be required to complete one maximal and sustained inspiratory effort from which the training is based on for that day.
  Interventions: Device: Test of Incremental Respiratory Endurance - IMT
- Threshold - IMT (Experimental): Subjects assigned to the Standard training regimen will receive a commonly used Threshold inspiratory muscle trainer. This device features a one-way spring-loaded valve at one end and a mouthpiece on the other through which subjects will be required to breathe in hard enough to overcome the resistance provided by the spring-loaded valve, allowing correct inspiration to happen. In other words, air flow is blocked until subjects generate sufficient inspiratory pressure to exceed the device pre-set pressure in cmH2O. The resistance will be set using the device's adjustable pressure setting which is fixed at 50% of the subject's MIP at the time of enrollment. The resistance will be readjusted as needed at week 4 to still reflect 50% of their inspiratory muscle strength at that time. Subjects will be coached to perform up to 36 breaths daily using the device. They will be also instructed to complete the training session within a 30-minute period.
  Interventions: Device: Threshold - IMT
- Sham IMT (Low resistence) (Sham Comparator): The Sham (Low Resistance) training regimen will use the same methods described above for the Standard IMT, except for the amount of resistance applied within the device. Subjects will receive a Threshold which has been set to its minimal resistance, which is 9 cmH2O. Again, subjects will be instructed to perform up to 36 breaths daily using the device within a 30-minute period.
  Interventions: Device: Sham IMT (Low resistence)

INTERVENTIONS:
Device: Test of Incremental Respiratory Endurance - IMT — The TIRE training regimen will involve the use of a tablet provided to assigned subjects with the training software installed and a PrO2® device through which they will train. The software allows subjects to track their inspiratory muscle performance via real-time graphic representations of their efforts as training progresses.
  Arms: Test of Incremental Respiratory Endurance - IMT
Device: Threshold - IMT — The Threshold incorporates a flow-independent one-way valve to ensure consistent resistance and features an adjustable specific pressure setting to be set based on MIP values of each subject.
  Arms: Threshold - IMT
Device: Sham IMT (Low resistence) — The Threshold incorporates a flow-independent one-way valve to ensure consistent resistance and features an adjustable specific pressure setting to be set based on MIP values of each subject.
  Arms: Sham IMT (Low resistence)

SUMMARY:
Subjects with chronic obstructive pulmonary disease (COPD) frequently develop considerable deterioration in exercise capacity in association with weakness and deconditioning of the respiratory muscles, which can be corrected with specific therapies. While pulmonary rehabilitation is a central component in the rather complex manangement of COPD, there is currently a lack of centers able to provide appropriate rehabilitation services in the Czech Republic. The main objective of this study will be to fully evaluate the utility of the Test of Incremental Respiratory Endurance (TIRE) as an at-home inspiratory muscle training method in subjects with COPD, while comparing the effectiveness of this novel training approach to the outcomes of more traditional ispiratory muscle training protocols.

This prospective, randomized controlled trial will include 2 treatment groups and 1 sham intervention group in a 1:1:1 ratio. All participants will undergo a certain type of IMT regardless of group assignment, which will be perfomed via two different devices. The trial will comprise of an 8-week at-home training period with remote supervision followed by 4 months of unsupervised, independent inspiratory muscle training. Study outcomes will include measures of inspiratory muscle strength and endurance, pulmonary function, COPD-specific symptomatology, functional exercise capacity, surrogate markers of mortality risk, mental health status and health-related quality of life of participants. While investigators acknowledge the value of standard inspiratory muscle training protocols which use Threshold devices, investigators believe that the TIRE training has the potential to provide additional clinical benefits since it is able to modulate all aspects of muscular performance, including strength, endurance and work capacity. Investigators hypothesize that, as a home-based stand-alone rehabilitative therapy, TIRE will be superior to standard IMT in improving COPD-related measures.

DETAILED DESCRIPTION:
Eligible participants will be randomly assigned to one of the following three distinct home-based IMT protocols: (1) TIRE, (2) Standard, and (3) Sham (i.e. Low Resistance). All subjects will undergo 8 weeks of daily unsupervised IMT using either a PrO2® device (Design Net, Smithfield, USA) or Threshold device at home. All training modalities require the subjects to be seated and wearing a nose clip while performing the required breaths. Subjects will be instructed on respective training procedures and complete first training session in the presence of a research team member upon enrollment. Regardless of training method, participants will be instructed to fill in diary cards at the end of each training session, in which participants document how many breaths were able to perform. This information will be later used for compliance assessment. Participants will be also provided with user guides developed by investigators research team with detailed instructions regarding equipment set-up, training protocol and contact information. In addition, subjects will receive weekly phone calls from week 0 to week 8 to encourage compliance and adherence to the study protocol, to address any subject questions or concerns, and to collect information regarding participants current symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* individuals over the age of 40
* clinical and functional diagnosis of COPD
* Global Initiative of Chronic Obstructive Lung Disease (GOLD) - stages I to IV
* evidence of inspiratory muscle weakness, defined as a MIP ≤ 80 cmH2O and a SMIP ≤ 427 PTU
* ability to operate a computer, tablet or smartphone
* clinical stability with no history of infections or exacerbation of respiratory symptoms for at least two months prior to study enrollment
* non-participation in exercise programs in the past 12 months.

Exclusion Criteria:

* subjects with history of lung surgery, lung cancer,
* any diagnosed cognitive (i.e. Mini Mental State Examination score < 24),
* orthopedic, neurological or neuromuscular disorders

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Sustained Maximal Inspiratory Pressure (SMIP) | Change from baseline to 8 weeks and 24 weeks
  The primary outcome measure will be SMIP, which will be obtained along with MIP and ID in every subject using the PrO2® device, an electronic pressure manometer which utilizes wireless technology to connect to a tablet containing the software of the Test of Incremental Respiratory Endurance.

SECONDARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Change from baseline to 8 weeks and 24 weeks
  MIP will be obtained from a maximal inspiratory effort from residual volume using the TIRE software and recorded in centimeters of water.
Inspiratory Duration (ID) | Change from baseline to 8 weeks and 24 weeks
  ID will be obtained from a maximal and sustained inspiratory effort using the TIRE software and recorded in seconds.

OTHER OUTCOMES:
Forced expiratory volume in the first second (FEV1) | Change from baseline to 8 weeks and 24 weeks
  FEV1 will be obtained from pulmonary function tests which comprise post-bronchodilator spirometry using SpiroScout® and whole-body plethysmography using the PowerCube® Body
Inspiratory capacity (IC) | Change from baseline to 8 weeks and 24 weeks
  IC will be obtained from pulmonary function tests which comprise post-bronchodilator spirometry using SpiroScout® and whole-body plethysmography using the PowerCube® Body
Forced vital capacity (FVC) | Change from baseline to 8 weeks and 24 weeks
  FVC will be obtained from pulmonary function tests which comprise post-bronchodilator spirometry using SpiroScout® and whole-body plethysmography using the PowerCube® Body
Six-minute Walk Test (6MWT) | Change from baseline to 8 weeks and 24 weeks
  Functional exercise capacity will be determined using the 6MWT. The best distance covered over a time of 6 minutes will be recorded in metres.
Modified Medical Research Council (mMRC) Dyspnea Scale | Change from baseline to 8 weeks and 24 weeks
  This scale ranges from zero to four, with higher scores indicating a greater degree of breathlessness.
Hospital Anxiety and Depression scale (HADS) | Change from baseline to 8 weeks and 24 weeks
  The questionnaire comprises seven questions for anxiety and seven questions for depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
St.George's Respiratory Questionnaire (SGRQ) | Change from baseline to 8 weeks and 24 weeks
  The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction. Scores range from 0 to 100, with higher scores indicating more limitations.
COPD Assessment Test (CAT) | Change from baseline to 8 weeks and 24 weeks
  This instrument that can quantify the impact of COPD on the patient's health. The CAT has a scoring range of 0-40. Higher scores denote a more severe impact of COPD.
Satisfaction - self-completed questionnaire | Change from baseline to 8 weeks and 24 weeks
  Subjects will be provided with a 5-item self-completed questionnaire developed by our research team that will measure their satisfaction with the intervention they received and the study in general. The items will be presented in the form of statements to which subjects will be asked to respond using a 1-5 Likert scale ("strongly agree", "agree", "not sure", "disagree", and strongly disagree").

CONTACTS AND LOCATIONS:
Overall Officials: Filip Dosbaba, PT, PhD, Study Director — University Hospital Brno, Czech Republic
Locations (1):
- University Hospital Brno, Brno, Czechia

REFERENCES:
- [Background] Formiga MF, Dosbaba F, Hartman M, Batalik L, Plutinsky M, Brat K, Ludka O, Cahalin LP. Novel versus Traditional Inspiratory Muscle Training Regimens as Home-Based, Stand-Alone Therapies in COPD: Protocol for a Randomized Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2020 Sep 11;15:2147-2155. doi: 10.2147/COPD.S266234. eCollection 2020. PMID 32982207
- See also: article link — https://doi.org/10.2147/COPD.S266234